CLINICAL TRIAL: NCT02292134
Title: Benefit of an Individual Protection Against Noise and Light on Sleep Quality in ICU Patients
Brief Title: Improving Sleep Quality in ICU Patients
Acronym: EARS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081115
Record Dates: First submitted 2013-11-21; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2013-11

CONDITIONS: Intensive Care Unit Patients
Keywords: Sleep quality; Sleep architecture; Intensive care unit; Light; Noise; Earplug; Sleep mask
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Ear Protective Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- earplug and sleep mask (Experimental)
  Interventions: Device: earplug and sleep mask
- control (No Intervention)

INTERVENTIONS:
Device: earplug and sleep mask — Individual protection against light and noise using earplugs and a sleep mask from 2 hrs to 8 hrs
  Arms: earplug and sleep mask

SUMMARY:
Sleep architecture is deeply altered in intensive care unit (ICU patients). Among factors involved in poor sleep quality are environmental factors, such as light and noise, which are an unavoidable consequence of cares.

The aim of the study is to evaluate the benefit of earplug and sleep mask on sleep architecture and quality in ICU patients.

DETAILED DESCRIPTION:
It is well demonstrated that sleep architecture is deeply altered in intensive care unit (ICU patients). The consequences of this alteration are multiple: neuropsychological complication such as delirium, long-term sequels such as post-traumatic stress disorders, alteration of the circadian fluctuation of various hormones with well demonstrated deleterious impact, alteration of the immune response that may promote nosocomial infections and, finally, a decrease of respiratory muscle endurance that may compromise weaning from mechanical ventilation.

Various mechanisms contribute to sleep alteration in ICU patients, including intrinsic factors linked to disease severity, factors related to therapies such as mechanical ventilation and sedation, and environmental factors. Among environmental factors, light and noise are an unavoidable consequence of cares that strongly contribute to sleep alteration in ICU patients. It is of notice that few studies have focused on strategies to protect ICU patients against noise and light such as the systematic use of earplug and sleep mask. Although the benefit of earplug and sleep mask on sleep quality has been demonstrated in healthy subjects submitted to an environment similar to ICU, it has never been evaluated in ICU patients.

The aim of the study is to evaluate the benefit of earplug and sleep mask (designated as "protective strategy) on sleep architecture and quality in ICU patients.

ELIGIBILITY:
Inclusion criteria :

* Admission in the ICU with expected duration of stay > 48hrs.
* Level of sedation < 4 on Ramsay scale.
* Interruption of sedation > 12 hrs
* Analgesia with a maximal dose of morphine < 0.01 mg/Kg/h
* Vasopressive therapy not exceeding 0.3 mg/Kg/min for epinephrine and 10 mg/Kg/min for dopamine.
* Informed consent by patients or next of kind.

Exclusion criteria :

* Known sleep disorder (apnea syndrome, narcolepsy, restless leg syndrome).
* Central nervous disease that might impact sleep architecture or the interpretation of EEG recordings.
* Severe liver encephalopathy (stage 3 or 4)
* Ongoing sepsis
* Pregnancy.
* Age < 18 yrs.
* No health insurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Duration of sleep stage 3 and 4 (polysomnography) | day 2
  Significant change of the duration of sleep stage 3 and 4 (polysomnography) in the "protective strategy group" (earplug and sleep mask) as compared to the control group (conventional strategy).

SECONDARY OUTCOMES:
Nocturnal awakenings (polysomnography) | Day 2
  in the "protective strategy group" (earplug and sleep mask) compared to the control group (conventional strategy).
Proportion of REM sleep (polysomnography) | Day 2
  in the "protective strategy group" (earplug and sleep mask) compared to the control group (conventional strategy).
Total sleep time (polysomnography) | Day 2
  in the "protective strategy group" (earplug and sleep mask) compared to the control group (conventional strategy).
Sleep time efficiency (polysomnography) | Day 2
  in the "protective strategy group" (earplug and sleep mask) compared to the control group (conventional strategy).
level of anxiety and depression (HAD scale) | At ICU discharge, an expected average of 3 weeks
  participants will be followed for the duration of ICU stay, a expected average of 3 weeks. comparison between the "protective strategy group" (earplug and sleep mask) and the control group (conventional strategy).
level of anxiety and depression (HAD scale) | At day 90
  comparison between the "protective strategy group" (earplug and sleep mask) and the control group (conventional strategy).
Incidence of posttraumatic stress disorder syndrome | At ICU discharge, an expected average of 3 weeks
  participants will be followed for the duration of ICU stay, a expected average of 3 weeks. comparison between the "protective strategy group" (earplug and sleep mask) and the control group (conventional strategy).
Incidence of posttraumatic stress disorder syndrome | At day 90
  comparison between the "protective strategy group" (earplug and sleep mask) and the control group (conventional strategy).

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit and Respiratory division ; Groupe hospitalier Pitie-Salpetriere and Universite Pierre et Marie Curie Paris 6, Paris, France

REFERENCES:
- [Derived] Demoule A, Carreira S, Lavault S, Pallanca O, Morawiec E, Mayaux J, Arnulf I, Similowski T. Impact of earplugs and eye mask on sleep in critically ill patients: a prospective randomized study. Crit Care. 2017 Nov 21;21(1):284. doi: 10.1186/s13054-017-1865-0. PMID 29157258